CLINICAL TRIAL: NCT05800860
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2b Trial With an Open-label Extension to Determine the Safety and Efficacy of GH001 in Patients With Treatment-resistant Depression
Brief Title: A Trial of GH001 in Patients With Treatment-resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GH Research Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GH001-TRD-201; 2022-000574-26 (EudraCT Number)
Record Dates: First submitted 2023-03-22; First posted 2023-04-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Treatment-resistant Depression
Keywords: Treatment-resistant depression; Major depressive disorder; Depression; GH001; 5-MeO-DMT; 5-methoxy-N,N-dimethyltryptamine; Mebufotenin
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Depression | interventions — Methoxydimethyltryptamines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GH001 - Part 1 (Experimental): GH001 is administered via inhalation, as an IDR consisting of up to 3 increasing doses of GH001 (6 mg, 12 mg, and 18 mg), on a single day. The second and third doses are only administered if the patient did not achieve intense psychoactive effects (a peak experience [PE]) at the previously administered dose.
  Interventions: Drug: GH001
- Placebo - Part 1 (Placebo Comparator): Placebo is administered via inhalation, as an IDR consisting of up to 3 doses of Placebo, on a single day. The second and third doses are only administered if the patient did not achieve intense psychoactive effects (a PE) at the previously administered dose.
  Interventions: Drug: Placebo
- Open-Label Extension (OLE) - Part 2 (Other): Patients can receive up to five GH001 IDRs as needed during the OLE based on the patient's clinical response.
  Interventions: Drug: GH001

INTERVENTIONS:
Drug: GH001 — GH001 administered via inhalation
  Other Names: 5-Methoxy-N,N-dimethyltryptamine; 5-MeO-DMT; Mebufotenin
  Arms: GH001 - Part 1; Open-Label Extension (OLE) - Part 2
Drug: Placebo — Placebo administered via inhalation
  Arms: Placebo - Part 1

SUMMARY:
The aim of this randomized, double-blind, placebo-controlled, phase 2b clinical trial is to investigate the safety and efficacy of GH001 (containing mebufotenin [5-methoxy-N,N-dimethyltryptamine; 5-MeO-DMT]) in patients with treatment-resistant depression (TRD). The study is comprised of a 7-day double-blind (DB) part (Part 1) and a 6-month open-label extension (OLE) part (Part 2). Patients will be randomized to receive GH001 or placebo in a 1:1 ratio. The primary endpoint is the mean change in the Montgomery-Åsberg Depression Rating Scale (MADRS) from baseline to Day 7.

DETAILED DESCRIPTION:
This is a phase 2b clinical trial in patients with TRD consisting of a 7-day randomized, placebo-controlled, DB Part 1 and a 6-month, single-arm, OLE Part 2. All patients who complete the DB Part 1 will directly transition into the OLE Part 2 on Day 7 of the DB Part 1.

In both parts, GH001 is administered as an individualized dosing regimen (IDR) consisting of up to 3 increasing doses of GH001 (6 mg, 12 mg, and 18 mg) on a single day, where the second and third doses are only administered if the patient did not achieve intense psychoactive effects (a peak experience [PE]) at the previously administered dose.

* In the DB Part 1, patients receive a single GH001 IDR or placebo IDR;
* In the OLE Part 2, patients can receive up to 5 GH001 IDRs as needed across 6 months, based on the patient's clinical response.

In both parts, an IDR clinic visit on Day (D)0 is followed by a telephone call on D1 and a clinic visit on D7 (±1 day).

The primary objective of this study is to determine the efficacy of a single day IDR of GH001 compared with placebo in improving depressive symptoms as assessed by the MADRS at the end of the 7-day DB Part 1.

Other efficacy objectives of this study are to assess the effects of the GH001 IDR on various measures of depression, anxiety and quality of life during the DB part and during the OLE. The safety of GH001 will also be assessed.

GH001 is an inhalation formulation of synthetic mebufotenin (5-MeO-DMT). The study drug is administered as an aerosol via pulmonary inhalation.

ELIGIBILITY:
Main Inclusion Criteria:

1. Is in the age range between 18 and 64 years (inclusive) at the time of informed consent;
2. Meets the trial criteria for TRD as assessed by a study psychiatrist:

   1. Meets the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) criteria for single-episode major depressive disorder (MDD) or recurrent MDD, without psychotic features confirmed by the Mini-International Neuropsychiatric Interview (MINI) with current episode duration of ≤2 years;
   2. The current major depressive episode must be deemed "valid" based upon the Massachusetts General Hospital State versus trait Assessability Face and Ecological validity Rule of 3Ps (MGH SAFER) criteria interview;
   3. Had nonresponse (≤25% improvement) to ≥2 and ≤5 oral antidepressant treatments administered during the current episode of depression.

Main Exclusion Criteria:

1. Has, based on history, psychiatric assessment, and evaluation of the MINI during the screening period, a first MDD episode after age 60, a current or prior diagnosis of a psychotic disorder, MDD, or other mood disorder with psychotic features, bipolar disorder, obsessive compulsive disorder, posttraumatic stress disorder, autism spectrum disorder, borderline personality disorder, schizophrenia, delusional disorder, paranoid personality disorder, schizoaffective disorder, clinically significant intellectual disability, antisocial personality disorder, schizotypal personality disorder, or any other psychiatric comorbidity that renders the patient unsuitable for the trial according to a study psychiatrist;
2. Has significant suicide risk;
3. Has 1 or more first degree relatives with a current or prior diagnosis of bipolar disorder, psychotic disorder, or other mood disorder (including MDD) with psychotic features;
4. Undergoing systematic psychotherapy that is planned to be modified or planning to initiate psychotherapy during the trial;
5. Has any current or past clinically significant condition that may interfere with the interpretation of the trial results, constitute a health risk for the patient, or that otherwise renders the patient unsuitable for the trial according to the investigator's judgement;
6. Fulfils criteria for DSM-5 alcohol or substance use disorder (excluding tobacco and caffeine use disorders) within the preceding 1 year, as assessed via the MINI;
7. Is taking antidepressants, antipsychotics, or any medication with monoamine oxidase inhibitors activity or takes or has taken other disallowed recent or concomitant treatments or it is anticipated that the patient will require treatment with at least 1 of the disallowed concomitant treatments during the trial;
8. Has previously experienced a significant adverse reaction to a hallucinogenic or psychedelic drug (e.g., psilocybin, Psilocybe spp. mushrooms, 5-MeO-DMT, DMT, ayahuasca, lysergic acid diethylamide, mescaline) according to the investigator's judgement.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Mean change in MADRS from Baseline to Day 7 | Baseline to Day 7
  The assessment is done with the MADRS, a diagnostic questionnaire with ten items for measuring the severity of depressive episodes in patients with mood disorders. A higher MADRS score indicates more severe depression, and each item is scored from 0 to 6. The overall score ranges from 0 to 60.

CONTACTS AND LOCATIONS:
Locations (11):
- Czechia (2):
  - Investigational site, Pilsen
  - Investigational site, Prague
- Germany (3):
  - Investigational Site, Dresden
  - Investigational Site, Frankfurt
  - Investigational Site, Münster
- Ireland (2):
  - Investigational site, Dublin
  - Investigational Site, Galway
- Investigational Site, Maastricht, Netherlands
- Investigational Site, Gdansk, Poland
- Spain (2):
  - Investigational Site, Barcelona
  - Investigational Site, Salamanca

IPD SHARING:
Plan to Share IPD: No